CLINICAL TRIAL: NCT02329223
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Omalizumab in Patients With Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite H1 Antihistamine Therapy
Brief Title: Study of Efficacy and Safety of Omalizumab in Refractory Chronic Spontaneous Urticaria Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025E2306
Record Dates: First submitted 2014-12-15; First posted 2014-12-31 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Spontaneous Uriticaria
Keywords: Chronic spontaneous uriticaria; Omalizumab
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omalizumab 300 mg (Experimental): Participants received omalizumab 300 mg subcutaneously every 4 weeks during the 12 week treatment period.
  Interventions: Biological: Omalizumab
- Omalizumab 150 mg (Experimental): Participants received omalizumab 150 mg subcutaneously every 4 weeks during the 12 week treatment period.
  Interventions: Biological: Omalizumab
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneously every 4 weeks during the 12 week treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Omalizumab — Omalizumab was supplied as a lyophilized, sterile powder in a single-use vial.
  Other Names: Xolair
  Arms: Omalizumab 150 mg; Omalizumab 300 mg
Other: Placebo — Placebo was supplied as a lyophilized, sterile powder in a single-use vial without study drug.
  Arms: Placebo

SUMMARY:
This was a Phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of omalizumab administered subcutaneously as an add-on therapy for the treatment of adolescent and adult participants 12 - 75 years who received the diagnosis of refractory chronic spontaneous uriticaria and who remained symptomatic despite standard-dosed non-sedating H1 antihistamine treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic spontaneous urticaria refractory to H1 antihistamine at the time of randomization
* Chronic spontaneous urticaria diagnosis for 6 months

Key Exclusion Criteria:

* Weight less than 20 kg
* Clearly defined underlying etiology for chronic urticaria other than chronic spontaneous urticaria
* Evidence of parasitic infection
* Any other skin diseases than chronic spontaneous urticaria with chronic itching
* Previous treatment with omalizumab
* Contraindications to diphenhydramine
* History of anaphylactic shock
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study
* History of hypersensitivity to omalizumab or to drugs of similar chemical classes
* Pregnant or nursing (lactating) women

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- Japan (23):
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kofu, Yamanashi
- South Korea (11):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to the 3 treatment groups in a 1:1:1 ratio.
Period: Overall Study
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Started | 73 | 71 | 74
Full Analysis Set | 73 | 70 | 74
Safety Set | 73 | 71 | 74
Completed | 72 | 68 | 68
Not Completed | 1 | 3 | 6
Not completed — Withdrawal by Subject | 1 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo | Total
Number analyzed (Participants) | 73 | 71 | 74 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (14.86) | 43.6 (12.24) | 42.5 (14.26) | 43.5 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 48 | 131
  Male | 33 | 28 | 26 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Itch Severity Score at Week 12
Description: The weekly itch severity score is a component of the Urticaria Activity Score 7 (UAS7) composite score. The UAS7 is a composite score of the number of wheals (hives) and the severity of the itch. The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score from baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: The Full Analysis Set (FAS) was analyzed. The FAS included all participants who were diagnosed with chronic spontaneous urticaria(CSU) and received the assigned study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Units on a scale | -10.22 (0.571) | -8.80 (0.591) | -6.51 (0.581)
Statistical Analysis 1: Comparison: Omalizumab 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Model with repeated measures(MMRM); Mean Difference (Net) = -3.70, 95% CI 2-sided [-5.310 to -2.098], Standard Error of Mean 0.815
Statistical Analysis 2: Comparison: Omalizumab 150 mg vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Model with repeated measures(MMRM); Mean Difference (Net) = -2.29, 95% CI 2-sided [-3.921 to -0.654], Standard Error of Mean 0.828

2. Secondary Outcome: Change From Baseline in the Urticaria Activity Score Over 7 Days (UAS7) at Week 12
Description: The UAS7 is a composite score of the number of wheals (hives) and the severity of the itch. The UAS7 is determined by the sum of the daily urticaria activity scores over 7 days and ranges from 0 to 42. The daily urticaria activity score is the average of the morning and evening urticaria activity scores and ranges from 0 to 6. The urticaria activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticaria activity scores over the 7 days prior to the first treatment. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: The Full Analysis Set (FAS) was analyzed. The FAS included all participants who were diagnosed with chronic spontaneous urticaria (CSU) and received the assigned study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Units on a scale | -22.44 (1.243) | -18.79 (1.288) | -13.90 (1.265)

3. Secondary Outcome: Change From Baseline in the Weekly Number of Hives Score at Week 12
Description: The weekly hives score is the sum of the daily hives scores over 7 days and ranges from 0 to 21. The number of hives is measured twice daily (morning and evening) on a scale of 0 (none) to 3 (> 12 hives per 12 hours). The daily hives score is the average of the morning and evening scores. The Baseline score is the sum of the daily hives scores over the 7 days prior to the first treatment. A higher score indicates more hives. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Units on a scale | -12.17 (0.742) | -10.04 (0.769) | -7.41 (0.756)

4. Secondary Outcome: Percentage of Participants With a UAS7 Score ≤ 6 at Week 12
Description: The UAS7 is a composite score of the number of wheals (hives) and the severity of the itch. The UAS7 is determined by the sum of the daily urticaria activity scores over 7 days and ranges from 0 to 42. The daily urticaria activity score is the average of the morning and evening urticaria activity scores and ranges from 0 to 6. The urticaria activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticaria activity scores over the 7 days prior to the first treatment. A higher urticaria activity score indicates more severe symptoms.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Percentage of participants | 57.5 | 42.9 | 18.9

5. Secondary Outcome: Change From Baseline in the Weekly Size of the Largest Hive Score at Week 12
Description: The weekly size of the largest hive score is the sum of the daily size of the largest hive scores over 7 days and ranges from 0 to 21. The daily size of the largest hive score is assessed twice daily (morning and evening) on a scale of 0 (none) to 3 (> 2.5 cm). The daily size of the largest hive score is the average of the morning and evening scores. The Baseline weekly size of the largest hive score is calculated over the 7 days prior to the first treatment. A higher score indicates larger hives. A negative change score from baseline indicates a reduction in hive size.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Units on a scale | -10.71 (0.684) | -9.30 (0.709) | -6.27 (0.696)

6. Secondary Outcome: Percentage of Weekly Itch Severity Score Minimally Important Difference (MID) Responders at Week 12
Description: Weekly itch severity score MID response is defined as a reduction from baseline in weekly itch severity score of ≥ 5 points.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Percentage of participants | 87.7 | 68.6 | 55.4

7. Secondary Outcome: Percentage of Complete Responders (UAS7 = 0) at Week 12
Description: Complete responders are defined as participants who achieved UAS7 = 0.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 74
Percentage of participants | 35.6 | 18.6 | 4.1

8. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a 10-item dermatology-specific health-related quality of life measure. Participants rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives on a scale of 0 (Not at all) to 3 (Very much). The overall DLQI is the sum of the responses to the 10 items and ranges from 0 to 30. A lower score indicates a better quality of life. A negative change score from baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: Only participants from the FAS, who were greater than age 16, were analyzed. The Full Analysis Set (FAS) was analyzed. The FAS included all participants who were diagnosed with chronic spontaneous urticaria (CSU) and received the assigned study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg | Placebo
Number analyzed (Participants) | 71 | 69 | 74
Units on a scale | -8.4 (0.52) | -7.2 (0.53) | -5.3 (0.52)

9. Secondary Outcome: Percentage of Participants With Production of Anti-omalizumab Antibody
Description: Serum samples were collected for anti-omalizumab antibody testing.
Time Frame: Week 24
Population: The safety analysis set, which included all participants who received their assigned study treatment, were considered for the analysis. Only participants, who had antibody results (conclusive or inconclusive), were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Omalizumab 300 mg | Omalizumab 150 mg
Number analyzed (Participants) | 68 | 64
Percentage of participants
  Conclusive results (n=64,63) | 0.0 | 0.0
  Inconclusive results (n=4,1) | NA — Results were inconclusive. | NA — Results were inconclusive.

ADVERSE EVENTS:
Time Frame: over 24 weeks following randomization
Groups:
- IGE025 300 mg: IGE025 300 mg
- IGE025 150 mg: IGE025 150 mg
- Placebo: Placebo
Arm/Group | IGE025 300 mg | IGE025 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/73 | 3/71 | 0/74
Other Adverse Events (participants affected / at risk) | 32/73 | 25/71 | 29/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 300 mg (N=73) | IGE025 150 mg (N=71) | Placebo (N=74)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 1 | 0
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 300 mg (N=73) | IGE025 150 mg (N=71) | Placebo (N=74)
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 2 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 1 | 2
CYSTITIS (Infections and infestations) | 0 | 2 | 0
FOLLICULITIS (Infections and infestations) | 1 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 9 | 7 | 12
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 2
PHARYNGITIS (Infections and infestations) | 3 | 3 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
HEADACHE (Nervous system disorders) | 3 | 3 | 5
MIGRAINE (Nervous system disorders) | 2 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 2 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 2
ACNE (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
CHRONIC SPONTANEOUS URTICARIA (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 5 | 3 | 2
MILIARIA (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
HYPERTENSION (Vascular disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.